CLINICAL TRIAL: NCT01802853
Title: Open Label, Randomized, 2 Way-crossover Study to Investigate the Absolute Bioavailability and Pharmacokinetics of RO6811135, Following Single Dose Administration by Subcutaneous and Intravenous Route in Healthy Subjects.
Brief Title: A Bioavailability and Pharmacokinetic Study of Subcutaneous and Intravenous RO6811135 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: BP28438; 2012-005773-31 (EudraCT Number)
Record Dates: First submitted 2013-02-28; First posted 2013-03-01 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer

ARMS (2):
- A: RO6811135 s.c. (Experimental)
  Interventions: Drug: RO6811135
- B: RO6811135 i.v. (Active Comparator)
  Interventions: Drug: RO6811135

INTERVENTIONS:
Drug: RO6811135 — Single subcutaneous dose
  Arms: A: RO6811135 s.c.
Drug: RO6811135 — Single intravenous dose
  Arms: B: RO6811135 i.v.

SUMMARY:
This open-label, randomized, 2-way crossover study will assess the absolute bioavailability and pharmacokinetics of RO6811135 in healthy male volunteers. Subjects will be randomized to one of the sequences AB or BA to receive single doses of subcutaneous (A) or intravenous (B) RO6811135, with a washout period of at least 7 days between dosing.

ELIGIBILITY:
Inclusion Criteria:

* Male healthy volunteers, 18-45 years of age inclusive
* Healthy as determined by screening assessments
* Body mass index (BMI) between 18-30 kg/m2

Exclusion Criteria:

* Any clinically relevant history or the presence of respiratory, renal, hepatic, gastrointestinal, hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological or connective tissue disease or diseases
* History of anaphylaxis or severe systemic hypersensitivity or allergic reactions
* Any history of alcohol and/or drug of abuse addiction during the past 5 years
* Smoking more than 5 cigarettes a day or the equivalent amount of tobacco
* Any clinically relevant abnormal test results prior to first dosing
* Positive for hepatitis B, hepatitis C or HIV infection
* Participation in an investigational drug or device study within 3 months prior to Day -1 of Period 1

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Absolute bioavailability of RO6811135 after subcutaneous administration: Area under the concentration-time curve (AUC) | 48 hours

SECONDARY OUTCOMES:
Safety: Incidence of adverse events | approximately 5 weeks
Pharmacodynamics: Fasting serum glucose/serum insulin | 48 hours
Nausea scale: Visual analogue scale | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Leeds, United Kingdom